CLINICAL TRIAL: NCT03600545
Title: Brain Fitness APP for Aging With a Healthy Brain and Detecting Cognitive Declines
Brief Title: Brain Fitness APP for Aging With a Healthy Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: AGE-WELL NCE Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2018:029
Record Dates: First submitted 2018-04-11; First posted 2018-07-26 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Memory Problems
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): 4 weeks daily practice of the brain exercises
  Interventions: Other: Brain Fitness App
- control (No Intervention): no brain exercises

INTERVENTIONS:
Other: Brain Fitness App — Brain exercises using an iPAD
  Arms: Active

SUMMARY:
Memory and cognitive declines are associated with normal brain aging but are also precursors to dementia, in particular the so called the pandemic of the century, Alzheimer's disease. While currently there is no cure or "vaccine" against dementia, there are hopes to delay the onset of the disease by living a brain-healthy life style. The proposed research offers a novel approach to prevent dementia and age-related cognitive disorders.

It is proposed to create a brain fitness APP for the aging population. The proposed APP is based on the premise of brain plasticity, and targets the brain functions that are declining with normal aging and dementia.

The proposed APP will be tested on a large population with statistical rigor (60 healthy individuals of age 65+ years and up to 30 individuals with cognitive impairment); the participants will be divided into an intervention group and a control group. We will analyze the logged performance of the participants, and assess their cognitive state with an independent test compared to a matched control group before and after the trial.

It is anticipated that the frequent use of the proposed APP will help to maintain a healthy brain as well as detecting the onset of a cognitive decline in aging population. In addition, its frequent use will slow and even reverse the progression of the cognition decline in individuals with mild cognitive impairment or dementia. The APP will have many different levels of difficulty so that it can be applied to a wide age range and conditions.

DETAILED DESCRIPTION:
The research is on the frequent use of our designed APP (for iPADs) that contains a series of our recently developed brain exercises that contains a series of our recently developed brain exercises, including orientation, associative memory, word-image association, recall memory, etc.

Participants will be randomly assigned to either Intervention or Control Arm. Participants of Intervention Arm must have access to an iPAD at least for the duration of the study.

Procedure for Intervention Arm The participants in Intervention Arm will have a training session (after obtaining their consent form) for the Brain Exercises. The Brain Fitness App will be downloaded into their iPAD and they will be instructed on how to use it. As mentioned in their consent form, they will commit themselves to play the games on a daily basis for (at least 5 days/week), twice/day, each session of minimum 15 minutes for a period of 4 consecutive weeks.

Procedure for Control Arm Participants of this arm will do nothing but will be assessed at baseline, 4 week and 8 weeks later. Their data will be used as the control data for comparison with the Intervention Arm data. All participants of this group, if interested, will be offered to practice the Brain Fitness App if they wish after their completion of this study (2 months period).

ELIGIBILITY:
Inclusion Criteria:

* MoCA ≥ 25
* Have no known or diagnosis of major depression, bipolar disorder, schizophrenia, mood disorder, Parkinson's disease, dementia of any type, or any other neurological degenerative disease.
* Capable of using an iPAD and access to Internet at home.
* Reading/writing fluency in English

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
The change in Wechsler Memory Scale (WMS IV) from baseline | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  This assessment has a total of 11 tests, out of which we will use its six primary tests that assess our target brain functions, comprised of 12 subtests (subsections): Logical Memory 1, Verbal Paired Associates 1, Faces 1, Family Pictures 1, Logical Memory 2, Verbal Paired Associates 2, Faces 2, Family Pictures 2, Verbal Paired Associates 2 Recognition, Logical Memory 2 Recognition, Letter-Number Sequencing and Spatial Span. They are classified into 3 major memory indexes: Immediate Memory, General Memory and Working Memory. The WMS test is being purchased online from the following link; they do not provide a softcopy.

SECONDARY OUTCOMES:
Change in Egocentric Spatial Orientation | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  This test is one of the PI's designs that has been in use since a few years ago. It is used for detecting the onset of Alzheimer's. In this test participants sit in a customized wheelchair and by waking the wheelchair they move within a virtual cubic building to reach a particular target room. They can do this test either using the laptop screen or in its immersive version wearing a goggle (Oculus Rift 2).
Change in MONTGOMERY ASBERG DEPRESSION RATING SCALE (MADRS) | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  The MADRS is a ten item rating scale for rating levels of depression. Each item is rated on a 7-point scale from 0 to 6, where 0 indicates absence of the symptom and 6 indicates extreme presence of the symptom. The time frame for the scale is the previous four weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada